CLINICAL TRIAL: NCT05585203
Title: Contingency Management for Recovery Oriented Activities at Recovery Houses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, David Ledgerwood, Associate Professor, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21-08-3875
Record Dates: First submitted 2022-10-05; First posted 2022-10-18 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Substance Use Disorders
Keywords: contingency management; Rural recovery houses
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design will be used. Half of the recovery houses residents will be randomly assigned to receive training in and to conduct contingency management. The other half will receive no additional training or interventions (usual care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency management (Experimental): In addition to receiving usual care at the recovery house, participants assigned to this arm will receive contingency management by trained recovery house staff in addition to their usual care. Contingency management sessions will be led by a trained recovery house staff member who is also a research participant in the study. Contingency management will occur once weekly for sessions of approximately 10-15 minute duration for up to 12 weeks. Participants will plan three recovery-oriented activities with the staff member each week, and upon verification of completion of the tasks, the resident participant can earn prize draws of varying monetary amounts.
  Interventions: Behavioral: Contingency management; Behavioral: Usual Care
- Usual Care (Active Comparator): Participants in this arm will receive usual care that they would normally receive at the recovery houses. Recovery houses are safe, healthy, family-like substance-free living environments that support individuals in recovery from addiction. Although recovery residences vary considerably, this form of housing benefits individuals in recovery by reinforcing a substance-free lifestyle and providing direct connections to other peers in recovery, mutual support groups and recovery support services.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Contingency management — The investigators will implement a prize-based contingency management protocol in which residents will complete three pre-planned recovery-oriented activities each week for a period of up to 12 weeks. Upon verified completion of the activities each week, participants may earn prize incentives through drawing from a prize fishbowl or spinning a virtual prize wheel.
  Prizes will be money added to a debit card. On the first week and individual has completed pre-planned activities, s/he can receive up to 1 draw per activity completed (3 total), and each week the number of prize draws per activity will escalate by 1. If a participant fails to complete any activities, he/she will not receive the draws for the uncompleted activities, and the prize draws would be reset to 1 in the next week. Participants can earn up to $75 in incentives in total.
  Arms: Contingency management
Behavioral: Usual Care — Participants in this arm will receive usual care that they would normally receive at the recovery houses. Recovery residences vary considerably, this form of housing benefits individuals in recovery by reinforcing a substance-free lifestyle and providing direct connections to other peers in recovery, mutual support groups and recovery support services.

SUMMARY:
In this study, the investigators will implement contingency management at rural recovery houses, where individuals with substance use disorders reside. Contingency management is a behavioral intervention in which participants receive incentives (rewards) when they complete planned tasks that are consistent with their recovery efforts. House staff members will also participate in this study and will be trained to provide contingency management to residents. The investigators will compare recovery houses that implement contingency management to matched houses that do not, and the main outcomes will be engagement in the planned activities and retention in the recovery houses. Participants will receive contingency management for up to 12 weeks and follow-up will occur 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older;
2. a resident of the recovery house; and
3. able to provide informed consent.

Exclusion Criteria:

1. expected to be discharged from the recovery house in the next two months;
2. experiencing uncontrolled mania, psychosis or suicidality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Treatment retention | Time until leaving the recovery home from study baseline up to one year
  Length of time (in days) a resident resides in the recovery house
Engagement in recovery-oriented activities | up to 12 week treatment
  Participants will engage in up to 3 planned recovery activities (noted on a tracking form)

SECONDARY OUTCOMES:
Treatment Satisfaction | Post-treatment (Week 12)
  Treatment Satisfaction Questionnaire (Scores range from 1 to 7 with higher scores reflecting greater satisfaction)
Quality of Life Assessment | Baseline, post-treatment (week 12) and 6-month follow up
  Self-report Quality of Life inventory (scores range from -3 to 3 with higher scores reflecting greater quality of life)
Self-Reported Health | Baseline, post-treatment (week 12) and 6-month follow up
  Short Form 36 (SF-36) is a brief measure of overall self-reported health. Scores range from 0 (maximum disability) to 100 (no disability)
Patient Health Questionnaire - 9 | Baseline, post-treatment (week 12) and 6-month follow up
  A measure of depression symptoms. Scores on the PHQ 9 range from 0 (no depression) to 27 (severe depression).
Substance Use | Baseline, weekly for 12 weeks, post-treatment (week 12) and 6-month follow up
  Urine drug screen of metabolites for cocaine, methamphetamine, barbiturates, opioids, cannabis, alcohol and benzodiazepines
Timeline Follow-back for substance use | Baseline, weekly for 12 weeks, post-treatment (week 12) and 6-month follow up
  Timeline Follow-back (TLFB) is a self-report, calendar-based measure of the frequency of substance use
Treatment Feasibility | Baseline
  Treatment Feasibility will assessed as the proportion of eligible participants who are willing to participate after initial screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University School of Medicine, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frisch, M.B., Cornell, J., Villanueva, M. & Retzlaff, P.J. (1992). Clinical validation of the quality of life inventory: A measure of life satisfaction for treatment planning and outcome assessment. Psychological Assessment, 4, 92-101.
- [Background] Novy, D.M., Nelson, D.V., Goodwin, J. & Rowzee, R.D. (1993). Psychometric comparability of the State-Trait Anxiety Inventory for different ethnic subpopulations. Psychological Assessment, 5, 343-349.
- [Background] Petry NM, Alessi SM, Ledgerwood DM. A randomized trial of contingency management delivered by community therapists. J Consult Clin Psychol. 2012 Apr;80(2):286-98. doi: 10.1037/a0026826. Epub 2012 Jan 16. PMID 22250852
- [Background] Petry NM, Alessi SM, Ledgerwood DM. Contingency management delivered by community therapists in outpatient settings. Drug Alcohol Depend. 2012 Apr 1;122(1-2):86-92. doi: 10.1016/j.drugalcdep.2011.09.015. Epub 2011 Oct 5. PMID 21981991
- [Background] Petry NM, Alessi SM, Ledgerwood DM, Sierra S. Psychometric properties of the contingency management competence scale. Drug Alcohol Depend. 2010 Jun 1;109(1-3):167-74. doi: 10.1016/j.drugalcdep.2009.12.027. Epub 2010 Feb 11. PMID 20149950
- [Background] Petry NM, Martin B, Finocche C. Contingency management in group treatment: a demonstration project in an HIV drop-in center. J Subst Abuse Treat. 2001 Sep;21(2):89-96. doi: 10.1016/s0740-5472(01)00184-2. PMID 11551737
- [Background] Rash CJ, Petry NM, Kirby KC, Martino S, Roll J, Stitzer ML. Identifying provider beliefs related to contingency management adoption using the contingency management beliefs questionnaire. Drug Alcohol Depend. 2012 Mar 1;121(3):205-12. doi: 10.1016/j.drugalcdep.2011.08.027. Epub 2011 Sep 16. PMID 21925807
- [Background] Shapiro, S.S. & Wilk, M.B. (1965). An analysis of variance test for normality (complete samples). Biometrika, 52.3/4, 591-611.
- [Background] Sobell, L.C., & Sobell, M.B. (1992). Timeline follow-back: A technique for assessing self-reported alcohol consumption. In R.Z. Litten and J.P. Allen (eds.), Measuring alcohol consumption: Psychosocial and biochemical methods (pp. 41-72). Totowa, NJ: Humana Press.
- [Background] Yi R, Johnson MW, Giordano LA, Landes RD, Badger GJ, Bickel WK. THE EFFECTS OF REDUCED CIGARETTE SMOKING ON DISCOUNTING FUTURE REWARDS: AN INITIAL EVALUATION. Psychol Rec. 2008 Spring;58(2):163-174. doi: 10.1007/BF03395609. PMID 23825867
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941